CLINICAL TRIAL: NCT02672865
Title: Adjuvant Hyperthermic Intraperitoneal Chemotherapy for Locally Advanced Gastric Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Maheswari Senthil, MD, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5150301
Record Dates: First submitted 2016-02-02; First posted 2016-02-03 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Locally Advanced Malignant Neoplasm; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- HIPEC (Experimental): The administration of hyperthermic intraperitoneal chemotherapy (HIPEC), using a warm solution of two chemotherapy medications (mitomycin and cisplatin) to bathe the internal surfaces of the abdomen in an attempt to kill any microscopic cancer cells that might be present on these surfaces.
  Interventions: Drug: Hyperthermic Intraperitoneal Chemotherapy (HIPEC)

INTERVENTIONS:
Drug: Hyperthermic Intraperitoneal Chemotherapy (HIPEC) — Hyperthermic intraperitoneal chemotherapy (HIPEC) is a procedure in which the internal parts of the abdomen are bathed in a warm solution of anti-cancer medications for 90 minutes.
  Other Names: HIPEC

SUMMARY:
The purpose of this study is to determine safety and feasibility of adjuvant hyperthermic intraperitoneal chemotherapy (HIPEC) with mitomycin and cisplatin in patients with locally advanced gastric cancer undergoing standard surgical resection. Patients will be treated with HIPEC using a single dose of mitomycin 15mg/m2 and cisplatin 50mg/m2 at 41-42 C for 90 minutes, during the definitive surgical resection for gastric cancer. HIPEC will be performed after resection but before anastomosis.

DETAILED DESCRIPTION:
Treatment Plan:

Patients undergoing definitive resection for gastric cancer and meeting the eligibility criteria will be treated with HIPEC using a single dose of Mitomycin 15mg/m2 and Cisplatin 50mg/m2 at 41-42 C for 90 minutes. HIPEC will be performed after resection but before anastomosis. Both Cisplatin and Mitomycin are commercially available chemotherapeutic agents and will be obtained as marketed drugs.

Outcome Measures:

Patients will be followed for 90 days following surgery. All postoperative complications will be recorded and graded according to the modified Clavien-Dindo classification.

Schedule for Follow Up:

Trial-related patient assessments will be performed daily while the patient remains in the hospital for postoperative care, and then during postoperative clinic visits. The final postoperative clinic visit for evaluation of study outcomes and complications should occur between postoperative days 90 and 95 to allow for a cumulative assessment of the patient's perioperative complications, if any.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-75 with biopsy-proven gastric adenocarcinoma
2. Tumor clinically staged T3 or T4 and/or nodes staged clinically positive
3. ECOG performance status < 2

Exclusion Criteria:

1. Distant metastases
2. Peritoneal carcinomatosis
3. Synchronous malignancy
4. Tumors at the gastroesophageal junction
5. Recurrent gastric adenocarcinoma
6. Creatinine >/= 1.5
7. Bilirubin >/= 2
8. INR >/= 2
9. Allergy to drugs included in the treatment plan
10. Pregnancy
11. Contraindication to major surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
Post Operative Complications | 90 days following surgery
  Patients will be followed for 90 days following surgery. Postoperative complications will be recorded and graded according to the modified Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Maheswari Senthil, MD, Principal Investigator — Loma Linda University Cancer Center
Locations (1):
- Loma Linda University Cancer Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Seshadri RA, Glehen O. Cytoreductive surgery and hyperthermic intraperitoneal chemotherapy in gastric cancer. World J Gastroenterol. 2016 Jan 21;22(3):1114-30. doi: 10.3748/wjg.v22.i3.1114. PMID 26811651
- [Result] Suo T, Mahteme H, Qin XY. Hyperthermic intraperitoneal chemotherapy for gastric and colorectal cancer in Mainland China. World J Gastroenterol. 2011 Feb 28;17(8):1071-5. doi: 10.3748/wjg.v17.i8.1071. PMID 21448361